CLINICAL TRIAL: NCT07388212
Title: Exploratory Study on LNP-mRNA Drugs Targeting CD19/BCMA for the Treatment of Relapsed and Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Liu, Professor, West China Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CD19/BCMA IIT for ADs
Record Dates: First submitted 2026-01-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD19/BCMA in vivo CAR-T, Escalation doses (Experimental)
  Interventions: Drug: CD19/BCMA in vivo CAR-T
- CD19/BCMA in vivo CAR-T, Extended doses (Experimental)
  Interventions: Drug: CD19/BCMA in vivo CAR-T

INTERVENTIONS:
Drug: CD19/BCMA in vivo CAR-T — CD19/BCMA in vivo CAR-T based on LNP-mRNA

SUMMARY:
Autoimmune diseases are a type of chronic disabling disease, characterized by the immune system incorrectly recognizing and attacking the body's own tissues, leading to tissue damage and organ dysfunction, seriously threatening life and health. Although there are various treatment methods currently available, there are still many limitations to immune related diseases that aim for long-term remission, and further research and breakthroughs are urgently needed.

Targeting and clearing B cells is one of the core strategies in the treatment of autoimmune diseases. Its mechanism mainly involves clearing abnormally activated B cells, reducing the production of autoantibodies, and regulating immune disorders. The therapy targeting CD19 has become an important research and development direction due to its ability to clear a wider range of B cell lineages (including plasma cells), which may achieve deeper levels of B cell depletion than CD20 targeted therapy. In addition, BCMA is highly expressed specifically on plasma cells, especially long-lived plasma cells, and is a key target for clearing the source of antibody production. Therefore, the CD19/BCMA dual target therapy aims to achieve more complete coverage of the antibody production pathway by simultaneously targeting B cells (and precursors) and plasma cells, which is expected to further improve the treatment response rate and achieve deeper and more persistent immune reset.

The advent of COVID-19 vaccine has brought LNP mRNA technology into the public's view. After years of development, it not only shines brilliantly in COVID-19 vaccine, but also is widely used in the treatment and exploration of cancer, rare diseases and other fields. The core of LNP mRNA technology targeting CD19/BCMA is to encapsulate the mRNA encoding specific proteins (such as anti-CD19/BCMA related proteins) in lipid nanoparticles and deliver them to the body through intravenous or intramuscular injection. This experimental drug is a messenger ribonucleic acid (mRNA) therapeutic drug based on the dual targets of CD19 and BCMA, formed by loading mRNA encoding CD19/BCMA receptor related proteins onto lipid nanoparticles (LNP) for injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of 18-70 years old (including threshold), gender not limited;
* 2. KPS score>60 points, life expectancy greater than 6 months;
* 3. Male and female patients of appropriate age must use reliable methods of contraception before entering the trial, during the research process until 30 days after discontinuation of medication; Reliable contraceptive methods will be determined by the primary researchers or designated personnel;
* 4. Those who can understand this experiment and have signed the informed consent form;
* 5. Before screening (at baseline), corresponding conditions should be met;
* 6. Disease related inclusion criteria (study participants must meet one of the following disease criteria): Indications for recurrent or refractory autoimmune diseases, including but not limited to systemic lupus erythematosus (SLE), etc.

Exclusion Criteria:

* 1. Study participants who are allergic or hypersensitive to any component of the investigational drug, including those who are allergic to messenger RNA (mRNA) vaccines or other RNA LNP products.
* 2. Merge any active infections that require antibiotic treatment and have not been controlled for at least one week prior to administration.
* 3. Accompanied by other uncontrolled malignant tumors.
* 4. History of cardiovascular disease within the first 6 months of screening: NYHA defined grade III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant heart diseases.
* 5. Positive for hepatitis B surface antigen (HBsAg); Or those who are positive for hepatitis B core antibody (HBcAb) and positive for hepatitis B virus (HBV) DNA or have a titer higher than the detection threshold; Individuals with positive hepatitis C virus (HCV) antibodies and HCV RNA positivity or titers above the detection threshold; Human immunodeficiency virus (HIV) antibody positive individuals; Cytomegalovirus (CMV) DNA positive or above the detection limit; Individuals who are positive for syphilis antigen or antibody.
* 6. Have received attenuated live vaccine or protein subunit vaccine within 30 days before the first study medication.
* 7. Women who are currently pregnant, breastfeeding, or planning to become pregnant.
* 8. The researchers believe that there are other situations that are not suitable for participating in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) and its incidence rate | Within 28 days after the initial treatment
Maxmum tolerated dose (MTD) or optimal biological dose (OBD) | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Preliminary efficacy evaluation: Objective Response Rate（ORR） | Through study completion, an average of 2 years
Preliminary efficacy evaluation: Duration of Response (DoR) | Through study completion, an average of 2 years